CLINICAL TRIAL: NCT00531791
Title: Effects of Fluticasone/Salmeterol (Advair®) in Outpatients With Chronic Obstructive Pulmonary Disease (COPD) Acute Exacerbation
Brief Title: Effects of Advair® in Outpatients With Chronic Obstructive Pulmonary Disease (COPD) Acute Exacerbation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Dre Julie Milot, Hôpital Laval
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCO-110754; CER 20222
Record Dates: First submitted 2007-09-17; First posted 2007-09-19 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; exacerbation; fluticasone; salmeterol; steroid
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: prednisone group
- 2 (Experimental)
  Interventions: Drug: Advair group

INTERVENTIONS:
Drug: prednisone group — Patients in the prednisone group will receive prednisone 40 mg per day with concomitant placebo diskus 2 inhalations twice a day for 10 days. All patients will receive oral antibiotics for 10 days, which will include moxifloxacin (Avelox®) 400 mg die or amoxicillin/clavulanate (Clavulin®) 875mg bid and short-acting bronchodilators (Ventolin®, Bricanyl®, Atrovent®) as needed.
  Arms: 1
Drug: Advair group — Patients in the second group will receive Advair® 50/500 ug 2 inhalations twice daily with placebo pills once a day for 10 days (twice the regular dosage). All patients will receive oral antibiotics for 10 days, which will include moxifloxacin (Avelox®) 400 mg die or amoxicillin/clavulanate (Clavulin®) 875mg bid and short-acting bronchodilators (Ventolin®, Bricanyl®, Atrovent®) as needed.
  Arms: 2

SUMMARY:
Short course of steroids in COPD exacerbation improves FEV1 and decreases the relapse rate. However, some concerns remain about using systemic steroids for all patients with acute exacerbation. Their short-term advantages may be outweighed by the occurrence of adverse side effects such as hyperglycemia, which is difficult to manage on an outpatient basis. In this context, the possibility of treating patients with COPD exacerbation with inhaled steroids having less systemic adverse effects is interesting. The objectives are to compare relapse rate, lung function, the severity of dyspnea and, systemic and sputum inflammatory markers in outpatients with acute COPD exacerbations treated with fluticasone/salmeterol (Advair®) or oral prednisone for 10 days. The hypothesis is that Advair® is as effective as prednisone in treatment of outpatients with COPD exacerbation. The primary endpoint is to determine if the relapse rate at one month is equivalent for both treatments. The secondary endpoints are to compare lung function and dyspnea score and, systemic and sputum inflammatory markers modulation after 10 days of both treatments. We will recruit 30 outpatients in each group from our COPD clinic. Patients will receive prednisone (40mg/day) with placebo diskus or Advair® 50/500ug 2 inhalations bid (twice the regular dose) with placebo pills for 10 days. All patients will receive antibiotics and short-acting bronchodilators as needed. We expect to demonstrate that the improvement of lung function, dyspnea, inflammatory markers and relapse rate are equivalent in both treatments suggesting that Advair® could be a good alternative to prednisone for patients with steroid-induced hyperglycemia.

DETAILED DESCRIPTION:
COPD exacerbations are a common cause of ill health, hospitalization and death. Once exacerbation symptoms are recognized, the current treatment consists of short course of oral steroids, antibiotics and increased bronchodilator intake. Systemic steroids are thought to reduce the inflammatory component of COPD exacerbation. A short course of steroid therapy improves FEV1 and decreases the relapse rate but most studies have been done on patients requiring hospitalization. Only few studies have described the role of steroids in the outpatients setting. However, some concerns remain about using systemic steroids for all patients with acute exacerbation. Their short-term advantages may be outweighed by the occurrence of adverse side effects such as hyperglycemia, which is difficult to manage on an outpatient basis. In this context, the possibility of treating patients with COPD exacerbation with inhaled steroids having less systemic adverse effects is interesting. In clinical trials, combination of corticosteroid with long-acting β2-adrenoceptor agonists (LABA) reduces airway inflammation, exacerbation rates, and improves lung function and health status of patients with stable moderate to severe COPD beyond that achieved by individual component therapy. Trials showed that nebulized steroid during acute COPD exacerbation requiring hospitalization is as effective as prednisone with less hyperglycemia. To our knowledge, no study has been conducted on the efficacy of combination treatment with inhaled steroid and LABA in the outpatient management of COPD exacerbation. Combination treatment could be a good alternative for patients with steroid contraindication and to reduce hospitalisation for uncontrolled hyperglycemia.

Primary objective: To compare relapse rates, lung function, the severity of dyspnea and, systemic and sputum inflammatory markers in outpatients with acute exacerbations of COPD treated with twice the regular dosage of Advair® or oral prednisone for 10 days.

Secondary objectives: To obtain preliminary data allowing sample size calculation for a larger similar clinical trial.

Hypothesis: Advair® is as effective as oral prednisone in treatment of outpatients with an acute COPD exacerbation.

Airway inflammation is a component of the pathophysiology of COPD exacerbation. Sputum from COPD-exacerbation patients has elevated inflammatory cells, TNF, IL-8 and RANTES levels compared to stable patients. Systemic steroid are thought to reduce the inflammatory component of COPD exacerbation. Appraisal of the current literature on glucocorticosteroids for acute COPD exacerbation show that a short course of systemic corticosteroid therapy improves spirometry and decreases the relapse rate but most studies using steroids for exacerbation have been done on patients requiring hospitalization, and only few have described the role of steroids in the outpatients setting. Two randomized controlled trials studied patients with acute COPD exacerbations not requiring hospitalization. Patients were assigned to receive oral prednisone for at least 9 days or placebo. The prednisone group showed a more rapid and significant improvement in forced expiratory volume at one second (FEV1). This therapy also resulted in fewer treatment failures and a trend toward more rapid improvement in dyspnea scale scores compared to placebo. However, despite proof of efficacy, some concerns remain about using systemic corticosteroid for all patients with acute exacerbation. Mainly because the short-term advantage may be outweighed by the occurrence of adverse side effects such as hyperglycemia, which is difficult to manage on outpatient basis and myopathy that can be observed even following a single oral dose of prednisolone. In this context, the possibility of treating patients with acute COPD exacerbation with inhaled corticosteroid having less systemic adverse effects is on particular interest.

Two trials have studied the effect of nebulized steroid during acute COPD exacerbation requiring hospitalization. Maltais et al. showed that 3 days of oral prednisone or nebulized budesonide significantly increased FEV1 compared to placebo. Compared with prednisone, nebulized budesonide was associated with a lesser occurrence of hyperglycemia, a potential advantage for diabetic patients with COPD. Recent studies have suggested long-acting b2-agonist as potential option in the treatment of acute exacerbation of COPD. It has been shown that salmeterol (up to 100 mcg) as formoterol (up to 48mcg) given over the same interval time induced an effective dose-dependent increase in FEV1, FVC and IC in patients with mild acute COPD exacerbation. Finally, the inhaled combination of salmeterol/fluticasone during 13 weeks in stable COPD patients showed a significant decrease in airway inflammation with decrease of lymphocytes, neutrophils, eosinophils and cells expressing genes for TNF and IFN. The main effect of inhaled corticosteroids is thought to be mediated through suppression of airway inflammation, while LABA are thought to work by inducing bronchodilation. However, there is emerging data to indicate that long-acting b2-adrenoceptor agonists may amplify the anti-inflammatory effects of corticosteroids by accelerating nuclear translocation of the glucocorticoid receptor complex, and enhancing transcription and expression of steroid-inducible genes in pro-inflammatory cells. These results suggest a role of the combination of long-acting b2-adrenoreceptor agonist and inhaled steroid in the inflammation observed in acute COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD
* history of 15 pack-years or more of cigarette smoking
* evidence of irreversible obstruction (FEV1<70% of predicted value, ratio FEV1/FVC<70%, and improvement of FEV1of less than 20% after bronchodilator in previous respiratory tests done when they were stable)

Exclusion Criteria:

* history of asthma or atopy
* need of being hospitalized
* use of oral or intravenous steroid within the preceding 30 days
* history of multiresistant bacterial infection (not applicable if absence of multi-resistant bacterial infection has been proved by a negative expectoration culture in the previous 6 months), bronchiectasis or recent COPD exacerbation (< 6 weeks) or diabetes.
* oxygen-dependant COPD patients or patients previously known with hypercapnia (PCO2>45 mmHg) at steady state
* use of high doses of Advair (more than 50/500 bid) or Symbicort (more than 12/400 bid)
* known cardiac arrhythmia such as atrial fibrillation, supraventricular tachycardia or paroxysmal auricular tachycardia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine, in patient with COPD presenting with an acute exacerbation that can be treated at home, if the relapse rate at one month is equivalent for both treatments. | September 2009

SECONDARY OUTCOMES:
To compare lung function and dyspnea score improvement 10 days post-treatment. | September 2009
To determine the systemic and sputum inflammatory marker modulations after 10 days of treatment and 30 days following the randomization. | September 2009

CONTACTS AND LOCATIONS:
Overall Officials: Julie Milot, MD PhD, Principal Investigator — Hôpital Laval, Institut universitaire de cardiologie et de pneumologie
Locations (1):
- Hôpital Laval, Institut universitaire de cardiologie et de pneumologie, Québec, Quebec, Canada